CLINICAL TRIAL: NCT05433025
Title: Safety and Treatment Effect of a Novel Device for Neck Pain in Active-duty Military Personnel With Forward Head Posture.
Brief Title: A Novel Device for Neck Pain in Active-duty Military Personnel With Forward Head Posture.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: The Geneva Foundation (Other); Walter Reed National Military Medical Center (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nathan Hogaboom, PhD, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WRNMMC-2021-0347
Record Dates: First submitted 2022-06-23; First posted 2022-06-27 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (Experimental): Cervigard Neck Collar, which is a device used to treat neck pain caused by forward head posture.
  Interventions: Device: Cervigard Neck Collar
- Waitlist Control (No Intervention): This group will receive no intervention for 6 weeks after enrollment. They will receive the device after 6 weeks.

INTERVENTIONS:
Device: Cervigard Neck Collar — A device used to treat neck pain caused by forward head posture
  Arms: Intervention

SUMMARY:
Neck pain is a common complaint among active duty military personnel, and can have tremendous impacts on quality of life and participation in duty-related activities. Treatments for spinal pain in military personnel are typically multimodal, relying upon physical therapy, pharmacological agents, spinal manipulation, and psychotherapy. However, there does not exist a wide body of evidence to support many of these treatments in active-duty military. The Cervigard neck collar was designed to treat posture-related neck pain with minimal effort and time required for treatment by the patient. However, this has yet to be tested experimentally. The objective of this study is to evaluate the treatment effect and safety of a novel device for the treatment of neck pain using self-reported pain and function measures, as well as objective radiological measures of cervical lordosis and head posture. Participants will be randomized to be fitted with and receive the Cervigard neck collar either immediately, or 6-weeks after being screened. Participants will complete neck pain and function questionnaires, and have cervical X-Rays collected at screening, treatment, 6 weeks, and 12 weeks (for the immediate group). Participants will be instructed to wear the collar every day for the duration of the trial. Self-reported neck pain and function measures will be collected, as well as cervical X-Rays, protocol adherence measures, and adverse events. The intervention is expected to reduce neck pain/discomfort, improve function, and improve cervical lordosis.

ELIGIBILITY:
Inclusion Criteria:

* DEERS Eligible
* Age 18 and 45 year old (inclusive)
* Neck pain duration ≥ 3 months without neurological signs and have been seen by a provider.
* Conventional treatments have not decreased neck pain
* Neck pain ≥ 4 on a 0-10 point numerical rating scale (0 = "no pain", 10 = "maximum pain")
* Forward head posture, indicated by forward placement of the head relative to the shoulders.

Exclusion Criteria:

* History of a tumor in the cervical spine and/or head/neck region within the past 6 months.
* Infection involving the cervical spine and/or head/neck region within the past 6 months.
* Generalized medical disorders that would weaken the vertebrae or other tissue structures within the cervical spine region.
* Fracture that is acute and/or still healing
* Spinal deformities (e.g. Fixed kyphosis, Ankylosing spondylosis)
* Medical and/or psychological condition that would preclude safe participation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Numerical Pain Rating Scale score | 6 weeks
  Neck pain intensity will be assessed using the Numerical Rating Scale. Subjects will be asked to rate their average pain during the past week using an 11-point scale (i.e. 0-10) anchored at the ends by "no pain" and "worst pain ever experienced."

SECONDARY OUTCOMES:
Change in Neck Disability Index scores | 6 weeks
  The Neck Disability Index is a disease-specific measure of neck pain-related sequelae. It includes 10 sections designed to capture different aspects of everyday life and how neck pain potentially affects those areas. Examples include personal care, lifting, headaches, concentration, work, and sleep.
Change in lordotic angle of the cervical spine | 6 weeks
  The angle of the curve of the cervical spine will be measured using a custom computer program in blinded and random fashion.
Change in head position | 6 weeks
  The position of the cranium relative to the 7th cervical vertebra will be measured using a custom computer program in blinded and random fashion.

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT05433025/ICF_000.pdf